CLINICAL TRIAL: NCT02288338
Title: CKD-391 in Healthy Volunteers to Investigate the Pharmacokinetic Drug Interaction Between Atorvastatin an Ezetimibe After Oral Administration
Brief Title: CKD-391 DDI : Atorvastatin and Ezetimibe in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 152DDI14016
Record Dates: First submitted 2014-10-30; First posted 2014-11-11 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
MeSH Terms: interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1(Lipitor®>Ezetrol®>Lipitor®, Ezetrol®) (Experimental): Three treatment
  1. atorvastatin calcium 40mg will be administration to healthy volunteers during 7days
  2. after 11days withdrawal period, ezetimibe 10mg will be administered to healthy volunteers during 7days
  3. after 11days withdrawal period, atorvastatin calcium 40mg and ezetimibe 10mg will be administered to healthy volunteers during 7days
  Interventions: Drug: 1 (Lipitor®); Drug: 1 (Ezetrol®); Drug: 1 (Lipitor®, Ezetrol®)
- 2(Ezetrol®>Lipitor®, Ezetrol®>Lipitor®) (Experimental): Three treatment
  1. ezetimibe 10mg will be administered to healthy volunteers during 7days
  2. after 11days withdrawal period, atorvastatin calcium 40mg and ezetimibe 10mg will be administered to healthy volunteers during 7days
  3. after 11days withdrawal period, atorvastatin calcium 40mg will be administered to healthy volunteers during 7days
  Interventions: Drug: 2 (Ezetrol®); Drug: 2(Lipitor®, Ezetrol®); Drug: 2 (Lipitor®)
- 3(Lipitor®, Ezetrol®>Lipitor®>Ezetrol®) (Experimental): Three treatment
  1. atorvastatin calcium 40mg and ezetimibe 10mg will be administered to healthy volunteers during 7days
  2. after 11days withdrawal period, atorvastatin calcium 40mg will be administered to healthy volunteers during 7days
  3. after 11days withdrawal period, ezetimibe 10mg will be administered to healthy volunteers during 7days
  Interventions: Drug: 3(Lipitor®, Ezetrol®); Drug: 3 (Lipitor®); Drug: 3 (Ezetrol®)
- 4(Lipitor®>Lipitor®, Ezetrol®>Ezetrol®) (Experimental): 1. atorvastatin calcium 40mg will be administered to healthy volunteers during 7days
  2. after 11days withdrawal period, atorvastatin calcium 40mg and ezetimibe 10mg will be administered to healthy volunteers during 7days
  3. after 11days withdrawal period, ezetimibe 10mg will be administered to healthy volunteers during 7days
  Interventions: Drug: 4 (Lipitor®); Drug: 4(Lipitor®, Ezetrol®); Drug: 4 (Ezetrol®)
- 5(Ezetrol®>Lipitor®>Lipitor®, Ezetrol®) (Experimental): 1. ezetimibe 10mg will be administered to healthy volunteers during 7days
  2. after 11days withdrawal period, atorvastatin calcium 40mg will be administered to healthy volunteers during 7days
  3. after 11days withdrawal period, atorvastatin calcium 40mg and ezetimibe 10mg will be administered to healthy volunteers during 7days
  Interventions: Drug: 5 (Ezetrol®); Drug: 5 (Lipitor®); Drug: 5 (Lipitor®, Ezetrol®)
- 6(Lipitor®, Ezetrol®>Ezetrol®>Lipitor®) (Experimental): 1. atorvastatin calcium 40mg and ezetimibe 10mg will be administered to healthy volunteers during 7days
  2. after 11days withdrawal period, ezetimibe 10mg will be administered to healthy volunteers during 7days
  3. after 11days withdrawal period, atorvastatin calcium 40mg will be administered to healthy volunteers during 7days
  Interventions: Drug: 6(Lipitor®, Ezetrol®); Drug: 6 (Ezetrol®); Drug: 6 (Lipitor®)

INTERVENTIONS:
Drug: 1 (Lipitor®) — atorvastatin calcium 40mg, Lipitor® 40mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg
  Arms: 1(Lipitor®>Ezetrol®>Lipitor®, Ezetrol®)
Drug: 1 (Ezetrol®) — After 11days withdrawal period, ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Ezetrol® 10mg
  Arms: 1(Lipitor®>Ezetrol®>Lipitor®, Ezetrol®)
Drug: 1 (Lipitor®, Ezetrol®) — After 11days withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg and ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg, Ezetrol® 10mg
  Arms: 1(Lipitor®>Ezetrol®>Lipitor®, Ezetrol®)
Drug: 2 (Ezetrol®) — ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Ezetrol® 10mg
  Arms: 2(Ezetrol®>Lipitor®, Ezetrol®>Lipitor®)
Drug: 2(Lipitor®, Ezetrol®) — After 11days withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg and ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg, Ezetrol® 10mg
  Arms: 2(Ezetrol®>Lipitor®, Ezetrol®>Lipitor®)
Drug: 2 (Lipitor®) — After 11day withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg
  Arms: 2(Ezetrol®>Lipitor®, Ezetrol®>Lipitor®)
Drug: 3(Lipitor®, Ezetrol®) — atorvastatin calcium 40mg, Lipitor® 40mg and ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg, Ezetrol® 10mg
  Arms: 3(Lipitor®, Ezetrol®>Lipitor®>Ezetrol®)
Drug: 3 (Lipitor®) — After 11day withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg
  Arms: 3(Lipitor®, Ezetrol®>Lipitor®>Ezetrol®)
Drug: 3 (Ezetrol®) — After 11day withdrawal period, ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Ezetrol® 10mg
  Arms: 3(Lipitor®, Ezetrol®>Lipitor®>Ezetrol®)
Drug: 4 (Lipitor®) — atorvastatin calcium 40mg, Lipitor® 40mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg
  Arms: 4(Lipitor®>Lipitor®, Ezetrol®>Ezetrol®)
Drug: 4(Lipitor®, Ezetrol®) — After 11days withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg and ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg, Ezetrol® 10mg
  Arms: 4(Lipitor®>Lipitor®, Ezetrol®>Ezetrol®)
Drug: 4 (Ezetrol®) — After 11day withdrawal period, ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Ezetrol® 10mg
  Arms: 4(Lipitor®>Lipitor®, Ezetrol®>Ezetrol®)
Drug: 5 (Ezetrol®) — ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Ezetrol® 10mg
  Arms: 5(Ezetrol®>Lipitor®>Lipitor®, Ezetrol®)
Drug: 5 (Lipitor®) — After 11day withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg
  Arms: 5(Ezetrol®>Lipitor®>Lipitor®, Ezetrol®)
Drug: 5 (Lipitor®, Ezetrol®) — After 11days withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg and ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg, Ezetrol® 10mg
  Arms: 5(Ezetrol®>Lipitor®>Lipitor®, Ezetrol®)
Drug: 6(Lipitor®, Ezetrol®) — atorvastatin calcium 40mg, Lipitor® 40mg and ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg, Ezetrol® 10mg
  Arms: 6(Lipitor®, Ezetrol®>Ezetrol®>Lipitor®)
Drug: 6 (Ezetrol®) — After 11days withdrawal period, ezetimibe 10mg, Ezetrol® 10mg will be administered to healthy volunteers during 7days
  Other Names: Ezetrol® 10mg
  Arms: 6(Lipitor®, Ezetrol®>Ezetrol®>Lipitor®)
Drug: 6 (Lipitor®) — After 11day withdrawal period, atorvastatin calcium 40mg, Lipitor® 40mg will be administered to healthy volunteers during 7days
  Other Names: Lipitor® 40mg
  Arms: 6(Lipitor®, Ezetrol®>Ezetrol®>Lipitor®)

SUMMARY:
A randomized open-label, multiple dose, three-treatment, three-period, six-sequence, crossover study to investigate the pharmacokinetic drug interaction between Atorvastatin and Ezetimibe after oral administration in healthy volunteers

DETAILED DESCRIPTION:
Outcome Measures

1. Primary endpoint AUCτ,ss, Cmax,ss of atorvastatin and free ezetimibe
2. Second endpoint 1) AUCinf,ss, Cavg,ss, %fluctuation, tmax,ss, t1/2, CL/Fss, Vd/Fss of atorvastatin and free ezetimibe 2) AUCτ,ss, AUCinf,ss, Cmax,ss, tmax,ss, t1/2, metabolic ratio of 2-hydroxy atorvastatin and free ezetimibe

ELIGIBILITY:
Inclusion Criteria:

1. Age Eligible for Study : 19 Years to 45 Years
2. If males, Body weight ≥ 55kg, If females, Body weight ≥ 50kg
3. BSA ≥ 18.5, <25
4. Accepts healthy volunteers
5. If female, Negative for pregnancy test at the screening and pre dose of Day 1
6. The subjects who agree with performing contraception during the study
7. The subjects who agreed with written informed consent

Exclusion Criteria:

1. The subjects with impaired hepatic function, renal function, nervous system etc.
2. The subjects have a gastrointestinal disease or surgery which can be effected in absorption of Investigational product
3. The subjects with high blood pressure or low blood pressure (Systolic blood pressure>150mmHg or <90mmHg, Diastolic blood pressure>100mmHg or <50mmHg
4. The subjects with abnormal Laboratory test (AST, ALT>1.25 fold of upper normal limit, Total bilirubin>1.5 fold of upper normal limit, CPK>2 fold of upper normal limit, Estimated Glomerular filtration rate<60mL/min/1.73m2 by Modification of Diet in Renal disease formula
5. The subjects have drug abuse history within 1year or Positive for urine drug test at screening
6. The subjects who took prescription only medicine whch can be effected in metabolism of Investigational product within 14days
7. The subjects who took over the counter drug whch can be effected in metabolism of Investigational product within 7days

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
Cmax,ss of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h

SECONDARY OUTCOMES:
AUCinf,ss of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
Cavg,ss of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
%fluctuation of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
tmax,ss of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
t1/2 of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
CL/Fss of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
Vd/Fss of atorvastatin and free ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
AUCτ,ss of 2-hydroxy atorvastatin and total ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
AUCinf,ss of 2-hydroxy atorvastatin and total ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
Cmax,ss of 2-hydroxy atorvastatin and total ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
tmax,ss of 2-hydroxy atorvastatin and total ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
t1/2 of 2-hydroxy atorvastatin and total ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h
metabolic ratio of 2-hydroxy atorvastatin and total ezetimibe | common : just before the IP administration of D5(D22, D39), D6(D23, D40)
  Atorvastatin single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48 h Ezetimibe single : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h Atorvastatin+Ezetimibe : just before the IP administration of D7(D24, D41) and after the IP administration 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 h

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D. M.D, Principal Investigator — Severance Hospital
Locations (1):
- ChongKunDang, Seoul, South Korea